CLINICAL TRIAL: NCT00336960
Title: Phase II Pilot Study of Pre-Operative Celecoxib (Celebrex) in Combination With Prolonged Venous Infusion 5FU and Radiation Therapy for Patients With Stage II/III Resectable Rectal Cancer
Brief Title: Celecoxib, Fluorouracil, and Radiation Therapy in Treating Patients With Stage II or Stage III Rectal Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0173; P50CA095103 (NIH); P30CA068485 (NIH); VICC-GI-0173; VICC-020031
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Celecoxib; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment intervention (Experimental)
  Interventions: Drug: celecoxib; Drug: fluorouracil; Procedure: conventional surgery; Radiation: radiation therapy; Procedure: tumor biopsy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: celecoxib — twice daily beginning 5 days prior to radiotherapy and continuing until completion of radiotherapy
Drug: fluorouracil — Patients receive concurrent fluorouracil IV continuously for 5 weeks.
Procedure: conventional surgery — 4-10 weeks after completion of chemoradiotherapy
Radiation: radiation therapy — Patients undergo radiotherapy 5 days a week for 5 weeks
Procedure: tumor biopsy — at baseline and then at the time of surgical resection
Other: laboratory biomarker analysis — blood and urine collected at baseline, 5 days after initiation of celecoxib, 7 days after initiation of celecoxib in combination with fluorouracil and radiotherapy, and at the time of surgical resection. specimens are evaluated for COX-2 expression, eicosanoid production, and gene and protein expression using immunohistochemistry, microarray, and mass spectrometry.

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Celecoxib may make tumor cells more sensitive to radiation therapy. Giving celecoxib together with fluorouracil and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving celecoxib together with fluorouracil and radiation therapy works in treating patients with stage II or stage III rectal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine cyclo-oxygenase-2 (COX-2) overexpression in patients with resectable stage II or III rectal cancer treated with neoadjuvant celecoxib, fluorouracil, and radiotherapy.
* Determine whether administration of celecoxib, a COX-2 inhibitor, results in changes in tumor (COX-2 overexpressing) levels of eicosanoids but not in the surrounding normal tissue.
* Determine if there is a greater change in protein and gene expression in post-treatment biopsies when compared to pretreatment biopsies that are greater for tumor (COX-2 overexpression) than in surrounding normal tissue.
* Determine whether patients who express the greatest degree of change in gene and protein expression are those most likely to respond to therapy.
* Assess the toxicities of concurrent treatment with celecoxib, fluorouracil, and radiotherapy.

OUTLINE: This is a pilot study.

Patients receive oral celecoxib twice daily beginning 5 days prior to radiotherapy and continuing until completion of radiotherapy. Patients undergo radiotherapy 5 days a week for 5 weeks. Patients also receive concurrent fluorouracil IV continuously for 5 weeks. Patients undergo radical resection 4-10 weeks after completion of chemoradiotherapy.

Patients undergo tumor biopsy at baseline and then at the time of surgical resection. Patients also undergo blood and urine collection at baseline, 5 days after initiation of celecoxib, 7 days after initiation of celecoxib in combination with fluorouracil and radiotherapy, and at the time of surgical resection. The specimens are evaluated for COX-2 expression, eicosanoid production, and gene and protein expression using immunohistochemistry, microarray, and mass spectrometry.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary adenocarcinoma of the rectum

  * Stage II or III disease
* Distal border of tumor must be at or below the peritoneal reflection

  * Distal border of the tumor must be within 12 cm of the anal verge by proctoscopic exam
* Tumor must be clinically resectable
* Transmural penetration beyond muscularis propria by transrectal ultrasound
* No high-grade obstruction
* No evidence of metastatic disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* WBC ≥ 4,000/mm³
* Platelet count ≥ 150,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious medical illness or psychiatric condition that would preclude study treatment
* No history of allergy to celecoxib or any other NSAIDs
* No history of allergy to sulfonamides
* No prior or concurrent malignancy except inactive noninvasive cervical carcinoma or skin cancer (excluding melanoma) or other cancer that has been disease free for ≥ 5 years

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the pelvis
* At least 7 days since prior and no other concurrent COX-2 inhibitors or nonsteroidal anti-inflammatory drugs (NSAIDs)
* No concurrent warfarin except low-dose warfarin (1 mg/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-07; Primary Completion 2004-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response rate | at time of surgery, day 5

SECONDARY OUTCOMES:
Complete resection rate | at time of surgery, day 5
Patterns of failure | during study, beginning day 5 forward
Survival | at time of death
Toxicity | 5 days before surgery & 5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee